CLINICAL TRIAL: NCT06030401
Title: Role Of Transthoracic Ultrasound in Predicting Post-extubation Distress During Successful Weaning
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Haredy Hassan Nafady, Resident physicion, Assiut University
Other Study IDs: Transthoracic US
Record Dates: First submitted 2023-08-09; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Transthoracic US

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transthoracic Ultrasound — Sonar of The Chest

SUMMARY:
-To Assess Value of Transthoracic Ultrasound In Predicting Post-extubation Distress in Respiratory ICU Using Ultrasound Parameters As Diaphragmatic Excursion ,Diaphragmatic,Diaphragmatic Thickness Fraction,Diaphragmatic Thickness.

DETAILED DESCRIPTION:
Establishing the correct time to extubate mechanically ventilated patients is a crucial issue in the critical care practice. Both premature and delayed extubation prolong the duration of mechanical ventilation and the intensive care unit (ICU) length of stay and increase morbidity and mortality. Therefore, accurate prediction of post-extubation distress and the early diagnosis of the causes responsible for failure of a trial of pressure support ventilation or a trial of totally unsupported respiration are of paramount importance to improve the outcome of mechanically ventilated patients in the ICU.

The Investigators hypothesized that the use of an integrative thoracic ultrasound assessment, encompassing bedside respiratory, and diaphragm sonographic data, could accurately predict post-extubation distress in patients who succeeded in a pressure support ventilation trial. In addition, The Investigators suggest that the use of appropriate analytical methods, that is, machine-learning methods, could permit the evaluation of the specific impact of respiratory and diaphragm sonographic data on the final estimation of a likelihood of post-extubation distress .

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 yrs. old who admitted to respiratory ICU and mechanically ventilated due to chest diseases and passed weaning trials

Exclusion Criteria:

* Pregnancy.
* Neuromuscular disorders.
* Psychiatric instability.
* Uncontrolled cardiovascular disease.
* Tracheostomy.
* patints with failed weaning trials.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: .Any Patient Has Successful Weaning Trial above18Years old in Respiratory ICU
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
post-extubation distress | "through study completion, an average of 3 year".
  Using Transthoracic US to measure Diaphragmatic Excursion and Diaphragmatic Thickness as Predictors of Postextubation Distress during Successful Weaning Trials.

SECONDARY OUTCOMES:
Evaluation of different factors that affect weaning outcome as diaphragmatic dysfunction,ventilator associated pneumonia,electrolyte disturbances and so on. | Doing Transthoracic US 48 hour after Starting of Mechanical Ventilation when Patient becomes Weanable during Weaning Trials,and 48 hour Postextubation Weaning and 48 hour postextubation.
  Looking on Diaphragmatic function And If There is any Ventilator Associated pneumonia And Electrolyte Disturbance

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Ahmad Ali, prof, Study Director — Respiratory ICU of Assiut University Hospital; Ali Abdelazeem Hassan, prof, Study Director — Respiratory ICU of Assiut University Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Follow Up of Intubated Patients During Weaning Trials Using Transthoracic US

REFERENCES:
- [Background] Frutos-Vivar F, Ferguson ND, Esteban A, Epstein SK, Arabi Y, Apezteguia C, Gonzalez M, Hill NS, Nava S, D'Empaire G, Anzueto A. Risk factors for extubation failure in patients following a successful spontaneous breathing trial. Chest. 2006 Dec;130(6):1664-71. doi: 10.1378/chest.130.6.1664. PMID 17166980
- [Result] Lichtenstein DA. Point-of-care ultrasound: Infection control in the intensive care unit. Crit Care Med. 2007 May;35(5 Suppl):S262-7. doi: 10.1097/01.CCM.0000260675.45549.12. PMID 17446786
- [Result] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Result] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Result] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Result] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2013 Mar 14;368(11):1068-9. doi: 10.1056/NEJMc1300398. No abstract available. PMID 23484845
- [Result] Epstein SK, Nevins ML, Chung J. Effect of unplanned extubation on outcome of mechanical ventilation. Am J Respir Crit Care Med. 2000 Jun;161(6):1912-6. doi: 10.1164/ajrccm.161.6.9908068. PMID 10852766
- [Result] Shen HN, Lin LY, Chen KY, Kuo PH, Yu CJ, Wu HD, Yang PC. Changes of heart rate variability during ventilator weaning. Chest. 2003 Apr;123(4):1222-8. doi: 10.1378/chest.123.4.1222. PMID 12684315
- [Result] Ueki J, De Bruin PF, Pride NB. In vivo assessment of diaphragm contraction by ultrasound in normal subjects. Thorax. 1995 Nov;50(11):1157-61. doi: 10.1136/thx.50.11.1157. PMID 8553271